CLINICAL TRIAL: NCT04148898
Title: A Randomized Phase II Trial of Osimertinib Alone or in Combination With Bevacizumab for EGFR- Mutant Non-small Cell Lung Cancer With Leptomeningeal Metastasis
Brief Title: Osimertinib With or Without Bevacizumab for EGFR- Mutant Non-small Cell Lung Cancer With Leptomeningeal Metastasis
Acronym: OWONBNSCLCLM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YC2019-S087
Record Dates: First submitted 2019-10-03; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Leptomeningeal Metastasis; Non-small Cell Lung Cancer; EGFR Activating Mutation
Keywords: leptomeningeal metastasis; non small cell lung cancer; EGFR Activating Mutation; Osimertinib; Bevacizumab
MeSH Terms: conditions — Meningeal Carcinomatosis; Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osimertinb group (Experimental): Osimertinib 80 mg oral daily
  Interventions: Drug: Osimertinib
- osimertinb combined with bevacizumab group (Experimental): Osimertinib 80 mg oral daily;
  .bevacizumab 7.5 mg/kg intravenous every 3 weeks
  Interventions: Drug: Osimertinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Osimertinib — Treatment of LM With osimertinb
  Other Names: AZD9291
Drug: Bevacizumab — Treatment of LM With osimertinb combined with bevacizumab
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb
  Arms: osimertinb combined with bevacizumab group

SUMMARY:
Leptomeningeal metastasis (LM) is a devastating and terminal complication of advanced non-small-cell lung cancer (NSCLC), especially in patients harboring epidermal growth factor receptor (EGFR) mutations. Osimertinib is an oral,third-generation, irreversible epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI) that selectively inhibits both EGFR-TKI-sensitizing and EGFR T790M resistance mutations .AURA I/II study and other preclinical study suggested that Osimertinib exhibited a better blood-brain barrier(BBB) penetration than the other EGFR-TKIs (gefitinib, erlotinib, or afatinib).The BLOOM 、AURA and FLURA study demonstrated that osimertinib showed encouraging activity and manageable tolerability in pretreated EGFR-mutant NSCLC patients with LM. Bevacizumab is a monoclonal antibody against vascular endothelial growth factor (VEGF). Animal study and autopsy specimens showed that VEGF is an essential factor in LM. Recently study showed EGFR-TKIs plus bevacizumab prolonged PFS and OS in patients with EGFR-mutant NSCLC and multiple brain mteastasis when compared with EGFR-TKIs alone. Howerver osimertinib combined with bevacizumab could benefit patients with LM from EGFR- mutant NSCLC remains undetermined. Therefore, the purpose of the study is to evaluate the safety and efficacy of osimertinib combined with bevacizumab for EGFR- mutant non-small cell lung cancer with leptomeningeal metastasis

DETAILED DESCRIPTION:
This is a randomized phase II clinical trial. The objective of the study is to assess the efficacy of osimertinib combined with bevacizumab for LM from EGFR- mutant NSCLC. Patients were randomized with equal allocation to 80 mg of oral Osimertinib daily alone or with 7.5 mg/kg of intravenous bevacizumab every 3 weeks. Study therapy continued until disease progression, unacceptable adverse event, or withdrawal of consent

ELIGIBILITY:
Inclusion Criteria:

* Age in 18-80 years
* Pathologically proven NSCLC
* EGFR mutation , the EGFR status was identified from primary lung tumors using the amplification refractory mutation system (ARMS) or next-generation sequencing (NGS) analysis.
* LM diagnosis was based on the detection of malignant cells in the CSF, the focal or diffuse enhancement of leptomeninges, and nerve roots or the ependymal surface on gadolinium-enhanced MRI .
* No severe abnormal liver and kidney function;
* No other severe chronic diseases;
* Signed informed consent form

Exclusion Criteria:

* Patients with the clinical manifestation of nervous system failure including severe encephalopathy, grade III-IV white matter lesions confirmed by imaging examination, moderate or severe coma, and glasgow coma score less than 9 points;
* Allergic to osimertinib or bevacizumab
* Any of the following: Pregnant women ;Nursing women ;Men or women of childbearing potential who are unwilling to employ adequate contraception
* History of myocardial infarction or other evidence of arterial thrombotic disease (angina), symptomatic congestive heart failure (New York Heart Association ≥ grade 2), unstable angina pectoris, or cardiac arrhythmia; Note: allowed only if patient has no evidence of active disease for at least 6 months prior to randomization;
* History of cerebral vascular accident (CVA) or transient ischemic attack (TIA)≤ 6 months prior to randomization
* History of bleeding diathesis or coagulopathy
* History of hemoptysis da≥ grade 2 (defined as bright red blood of at least 2.5 mL) ≤3 months prior to randomization
* Leukocytes below 2*10^9/L, neutrophils below 1*10^9/L; platelets below 50*10^9/L;
* Had major surgery within 60 days;
* History of arteriovenous thrombosis
* Gastrointestinal perforator in the past 6 months
* Inadequately controlled hypertension (systolic blood pressure of > 150 mmHg or diastolic pressure > 100 mmHg on anti-hypertensive medications); Note: history of hypertensive crisis or hypertensive encephalopathy not allowed
* Grade 4 proteinuria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free | Every 6 weeks, up to 2 years,
  iPFS (Time from LM diagnosis to the first documentation of intracranial lesion progression or death with documented intracranial pro- gression,)
Objective Response Rate | Every 6 weeks, up to 2 years
  ORR, proportion of patients with a best overall response of complete response or partial response (CR+PR)

SECONDARY OUTCOMES:
LM Overall survival | Every 3 weeks, up to 5 years,
  LM-OS defined as time from LM diagnosis to death due to any cause or last follow-up
progression-free survival | Every 6 weeks, up to 2 years,
  Proportion of patients progression-free by investigator assessment per RECIST v1.1
adverse events | Every 3 weeks, up to 2 years,
  Number of patients with adverse events (AEs) as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Liu Anwen, Phd, Study Director — Second Affiliated Hospital of Nanchang University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai Z, Liu Q. Understanding the Global Cancer Statistics 2018: implications for cancer control. Sci China Life Sci. 2021 Jun;64(6):1017-1020. doi: 10.1007/s11427-019-9816-1. Epub 2019 Aug 26. No abstract available. PMID 31463738
- [Background] Liao BC, Lee JH, Lin CC, Chen YF, Chang CH, Ho CC, Shih JY, Yu CJ, Yang JC. Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors for Non-Small-Cell Lung Cancer Patients with Leptomeningeal Carcinomatosis. J Thorac Oncol. 2015 Dec;10(12):1754-61. doi: 10.1097/JTO.0000000000000669. PMID 26334749
- [Background] Zhou Q, Song Y, Zhang X, Chen GY, Zhong DS, Yu Z, Yu P, Zhang YP, Chen JH, Hu Y, Feng GS, Song X, Shi Q, Yang LL, Zhang PH, Wu YL. A multicenter survey of first-line treatment patterns and gene aberration test status of patients with unresectable Stage IIIB/IV nonsquamous non-small cell lung cancer in China (CTONG 1506). BMC Cancer. 2017 Jul 3;17(1):462. doi: 10.1186/s12885-017-3451-x. PMID 28673332
- [Background] Wu YL, Zhao Q, Deng L, Zhang Y, Zhou XJ, Li YY, Yu M, Zhou L, Zou BW, Lu Y, Liu YM. Leptomeningeal metastasis after effective first-generation EGFR TKI treatment of advanced non-small cell lung cancer. Lung Cancer. 2019 Jan;127:1-5. doi: 10.1016/j.lungcan.2018.11.022. Epub 2018 Nov 20. PMID 30642536
- [Background] Cheng H, Perez-Soler R. Leptomeningeal metastases in non-small-cell lung cancer. Lancet Oncol. 2018 Jan;19(1):e43-e55. doi: 10.1016/S1470-2045(17)30689-7. PMID 29304362
- [Background] Reijneveld JC, Taphoorn MJ, Kerckhaert OA, Drixler TA, Boogerd W, Voest EE. Angiostatin prolongs the survival of mice with leptomeningeal metastases. Eur J Clin Invest. 2003 Jan;33(1):76-81. doi: 10.1046/j.1365-2362.2003.01056.x. PMID 12492456
- [Background] Ballard P, Yates JW, Yang Z, Kim DW, Yang JC, Cantarini M, Pickup K, Jordan A, Hickey M, Grist M, Box M, Johnstrom P, Varnas K, Malmquist J, Thress KS, Janne PA, Cross D. Preclinical Comparison of Osimertinib with Other EGFR-TKIs in EGFR-Mutant NSCLC Brain Metastases Models, and Early Evidence of Clinical Brain Metastases Activity. Clin Cancer Res. 2016 Oct 15;22(20):5130-5140. doi: 10.1158/1078-0432.CCR-16-0399. Epub 2016 Jul 19. PMID 27435396
- [Background] Jiang T, Chu Q, Wang H, Zhou F, Gao G, Chen X, Li X, Zhao C, Xu Q, Li W, Wu F, Xiong A, Zhao J, Xu Y, Su C, Ren S, Zhou C, Hirsch FR. EGFR-TKIs plus local therapy demonstrated survival benefit than EGFR-TKIs alone in EGFR-mutant NSCLC patients with oligometastatic or oligoprogressive liver metastases. Int J Cancer. 2019 May 15;144(10):2605-2612. doi: 10.1002/ijc.31962. Epub 2018 Dec 8. PMID 30387880
- [Background] Wu YL, Ahn MJ, Garassino MC, Han JY, Katakami N, Kim HR, Hodge R, Kaur P, Brown AP, Ghiorghiu D, Papadimitrakopoulou VA, Mok TSK. CNS Efficacy of Osimertinib in Patients With T790M-Positive Advanced Non-Small-Cell Lung Cancer: Data From a Randomized Phase III Trial (AURA3). J Clin Oncol. 2018 Sep 10;36(26):2702-2709. doi: 10.1200/JCO.2018.77.9363. Epub 2018 Jul 30. PMID 30059262
- [Background] Le Rhun E, Weller M, Brandsma D, Van den Bent M, de Azambuja E, Henriksson R, Boulanger T, Peters S, Watts C, Wick W, Wesseling P, Ruda R, Preusser M; EANO Executive Board and ESMO Guidelines Committee. EANO-ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up of patients with leptomeningeal metastasis from solid tumours. Ann Oncol. 2017 Jul 1;28(suppl_4):iv84-iv99. doi: 10.1093/annonc/mdx221. No abstract available. PMID 28881917